CLINICAL TRIAL: NCT02946463
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study of ALXN1210 Versus Eculizumab in Complement Inhibitor-Naïve Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: ALXN1210 (Ravulizumab) Versus Eculizumab in Complement Inhibitor Treatment-Naïve Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-301; 2016-002025-11
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab; eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental)
  Interventions: Biological: Ravulizumab
- Eculizumab (Active Comparator)
  Interventions: Biological: Ravulizumab; Biological: Eculizumab

INTERVENTIONS:
Biological: Ravulizumab — All treatments were given as intravenous (IV) infusions. For participants weighing ≥40 to <60 kilogram (kg): 2400 mg was given as a single loading dose, followed by 3000 mg as maintenance dose. For participants weighing ≥60 to <100 kg: 2700 mg was given as a loading dose, followed by 3300 mg as maintenance dose. For participants weighing ≥100 kg: 3000 mg was given as a loading dose, followed by 3600 mg as maintenance dose.
Biological: Eculizumab — All treatments were given as IV infusions. Participants were administered induction doses of 600 mg followed by maintenance doses of 900 mg.
  Arms: Eculizumab

SUMMARY:
The primary purpose of this study was to assess the noninferiority of ravulizumab compared to eculizumab in adult participants with PNH who had never been treated with a complement inhibitor (treatment-naïve).

DETAILED DESCRIPTION:
The study consisted of a 4-week screening period and a 26-week randomized treatment period (Primary Evaluation Period). After completion of the 26-week Primary Evaluation Period, all participants had the opportunity to enter the Extension Period, wherein participants will receive ravulizumab for up to 5 years.

ELIGIBILITY:
Criteria For Patient Cohort Originally Enrolled in ALXN1210-PNH-301 Study: Inclusion Criteria: 1. Male or female ≥18 years of age. 2. PNH diagnosis confirmed by documented by high-sensitivity flow cytometry. 3. Presence of 1 or more of the following PNH-related signs or symptoms within 3 months of screening: fatigue, hemoglobinuria, abdominal pain, shortness of breath (dyspnea), anemia (hemoglobin <10 gram/deciliter), history of a major adverse vascular event (including thrombosis), dysphagia, or erectile dysfunction; or history of packed red blood cells (pRBC) transfusion due to PNH. 4. Lactate dehydrogenase (LDH) level ≥1.5 times the upper limit of normal at screening. 5. Documented meningococcal vaccination not more than 3 years prior to, or at the time of, initiating study treatment. 6. Female participants of childbearing potential must use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab. 7. Willing and able to give written informed consent and comply with study visit schedule. Exclusion Criteria: 1. Treatment with a complement inhibitor at any time. 2. History of bone marrow transplantation. 3. Body weight <40 kg. 4. Females who are pregnant, breastfeeding, or who have a positive pregnancy test at screening or Day 1. 5. Participation in another interventional clinical study or use of any experimental therapy within 30 days before initiation of study drug on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater. 6. History of or ongoing major cardiac, pulmonary, renal, endocrine, or hepatic disease that, in the opinion of the investigator or sponsor, would preclude participation. 7. Unstable medical conditions (for example, myocardial ischemia, active gastrointestinal bleed, severe congestive heart failure, anticipated need for major surgery within 6 months of randomization, coexisting chronic anemia unrelated to PNH). Eligibility Criteria For Roll-over Cohort: 1. All participants regardless of age, who are currently receiving ALXN1210 IV in an ongoing ALXN1210 study in patients with PNH 2. Participants must be willing and able to give written informed consent and to comply with all Extension study visits and procedures, including the use of any data collection device(s) to directly record patient data 3. Females of childbearing potential and male patients with female partners of childbearing potential must use highly effective contraception continuing until at least 8 months after the last dose of ravulizumab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (104):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Whittier, California
  - Research Site, Fort Worth, Texas
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
- Research Site, Perth, Australia
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Hasselt
  - Research Site, Leuven
- Brazil (3):
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
- Czechia (2):
  - Research Site, Pilsen
  - Research Site, Prague
- Research Site, Tallinn, Estonia
- France (6):
  - Research Site, Limoges
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rennes
- Germany (3):
  - Research Site, Aachen
  - Research Site, Essen
  - Research Site, Ulm
- Italy (5):
  - Research Site, Ascoli Piceno
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Vicenza
- Japan (22):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hamamatsu
  - Research Site, Kanazawa
  - Research Site, Kitakyusyu-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumamoto
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Ogaki-shi
  - Research Site, Okayama
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Shimotsuke-shi
  - Research Site, Shinjuku-ku
  - Research Site, Suita
  - Research Site, Tokorozawa-shi
  - Research Site, Tokyo
  - Research Site, Toyoake-shi
  - Research Site, Tsukuba
  - Research Site, Wakayama
- Malaysia (7):
  - Research Site, George
  - Research Site, Johor Bahru
  - Research Site, Kota Bharu
  - Research Site, Kota Kinabalu
  - Research Site, Kuching
  - Research Site, Miri
  - Research Site, Sibu
- Research Site, Monterrey, Mexico
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Russia (13):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ufa
- Research Site, Belgrade, Serbia
- Research Site, Singapore, Singapore
- South Korea (10):
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, JinJoo
  - Research Site, Junggu
  - Research Site, Seoul
  - Research Site, Songpa-gu
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (2):
  - Research Site, Madrid
  - Research Site, Majadahonda
- Research Site, Uppsala, Sweden
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Hualien City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Songkhla
- Research Site, Eskişehir, Turkey (Türkiye)
- United Kingdom (3):
  - Research Site, Airdrie
  - Research Site, Leeds
  - Research Site, London

REFERENCES:
- [Background] Lee JW, Sicre de Fontbrune F, Wong Lee Lee L, Pessoa V, Gualandro S, Fureder W, Ptushkin V, Rottinghaus ST, Volles L, Shafner L, Aguzzi R, Pradhan R, Schrezenmeier H, Hill A. Ravulizumab (ALXN1210) vs eculizumab in adult patients with PNH naive to complement inhibitors: the 301 study. Blood. 2019 Feb 7;133(6):530-539. doi: 10.1182/blood-2018-09-876136. Epub 2018 Dec 3. PMID 30510080
- [Derived] Schrezenmeier H, Kulasekararaj A, Mitchell L, de Latour RP, Devos T, Okamoto S, Wells R, Popoff E, Cheung A, Wang A, Tomazos I, Patel Y, Lee JW. Predictors for improvement in patient-reported outcomes: post hoc analysis of a phase 3 randomized, open-label study of eculizumab and ravulizumab in complement inhibitor-naive patients with paroxysmal nocturnal hemoglobinuria. Ann Hematol. 2024 Jan;103(1):5-15. doi: 10.1007/s00277-023-05483-0. Epub 2023 Oct 7. PMID 37804344
- [Derived] Schwartz CE, Stark RB, Borowiec K, Nolte S, Myren KJ. Norm-based comparison of the quality-of-life impact of ravulizumab and eculizumab in paroxysmal nocturnal hemoglobinuria. Orphanet J Rare Dis. 2021 Sep 15;16(1):389. doi: 10.1186/s13023-021-02016-8. PMID 34526067
- [Derived] Schrezenmeier H, Kulasekararaj A, Mitchell L, Sicre de Fontbrune F, Devos T, Okamoto S, Wells R, Rottinghaus ST, Liu P, Ortiz S, Lee JW, Socie G. One-year efficacy and safety of ravulizumab in adults with paroxysmal nocturnal hemoglobinuria naive to complement inhibitor therapy: open-label extension of a randomized study. Ther Adv Hematol. 2020 Oct 24;11:2040620720966137. doi: 10.1177/2040620720966137. eCollection 2020. PMID 33178408
- [Derived] Ishiyama K, Nakao S, Usuki K, Yonemura Y, Ikezoe T, Uchiyama M, Mori Y, Fukuda T, Okada M, Fujiwara SI, Noji H, Rottinghaus S, Aguzzi R, Yokosawa J, Nishimura JI, Kanakura Y, Okamoto S. Results from multinational phase 3 studies of ravulizumab (ALXN1210) versus eculizumab in adults with paroxysmal nocturnal hemoglobinuria: subgroup analysis of Japanese patients. Int J Hematol. 2020 Oct;112(4):466-476. doi: 10.1007/s12185-020-02934-6. Epub 2020 Aug 31. PMID 32869125
- [Derived] Brodsky RA, Peffault de Latour R, Rottinghaus ST, Roth A, Risitano AM, Weitz IC, Hillmen P, Maciejewski JP, Szer J, Lee JW, Kulasekararaj AG, Volles L, Damokosh AI, Ortiz S, Shafner L, Liu P, Hill A, Schrezenmeier H. Characterization of breakthrough hemolysis events observed in the phase 3 randomized studies of ravulizumab versus eculizumab in adults with paroxysmal nocturnal hemoglobinuria. Haematologica. 2021 Jan 1;106(1):230-237. doi: 10.3324/haematol.2019.236877. PMID 31949012
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-PNH-301&attachmentIdentifier=dadc661d-a7a3-4ea9-8bde-01f258a0442b&fileName=ALXN1210-PNH-301-CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 adult and 2 pediatric participants rolled over from other Alexion ongoing studies of ravulizumab intravenous in participants with PNH into the extension period of this study and received weight-based doses of ravulizumab until end of study.
Pre-assignment Details: Participants were stratified into 6 groups based on transfusion history and LDH screening levels. Stratified participants were then randomly assigned in a 1:1 ratio to receive either ravulizumab or eculizumab in the 26-week Primary Evaluation Period.
Groups:
- Ravulizumab/Ravulizumab: Participants received weight-based doses of ravulizumab ranging from 2400 to 3000 mg on Day 1. Thereafter, weight-based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Day 15 and every 8 weeks thereafter for 26 weeks. After completion of the Primary Evaluation Period, all participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 5 years.
- Eculizumab/Ravulizumab: Participants received 600 mg of eculizumab on Days 1, 8, 15, and 22, followed by 900 mg of eculizumab on Day 29 and every 2 weeks thereafter for 26 weeks. After completion of the Primary Evaluation Period, all participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 5 years.
- Roll-Over Cohort: Ravulizumab - Adults; Roll-Over Cohort: Ravulizumab - Pediatrics: Participants in this group rolled over from other ongoing studies of ravulizumab intravenous in participants with PNH into the extension period of this study and received weight-based doses of ravulizumab for up to 5 years.
Period: Primary Evaluation Period
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab | Roll-Over Cohort: Ravulizumab - Adults | Roll-Over Cohort: Ravulizumab - Pediatrics
Started | 125 | 121 | 0 | 0
Received at Least 1 Dose of Study Drug | 125 | 121 | 0 | 0
Completed | 125 | 119 | 0 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Extension Period
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab | Roll-Over Cohort: Ravulizumab - Adults | Roll-Over Cohort: Ravulizumab - Pediatrics
Started (1 participant did not enter the Extension Period.) | 124 | 119 | 24 | 2
Received at Least 1 Dose of Ravulizumab | 124 | 119 | 24 | 2
Completed | 108 | 102 | 22 | 2
Not Completed | 16 | 17 | 2 | 0
Not completed — Death | 4 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 0 | 0
Not completed — Other than specified | 2 | 3 | 2 | 0
Not completed — Physician Decision | 1 | 4 | 0 | 0
Not completed — Pregnancy | 3 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab | Roll-Over Cohort: Ravulizumab - Adults | Roll-Over Cohort: Ravulizumab - Pediatrics | Total
Number analyzed (Participants) | 125 | 121 | 24 | 2 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 2 | 2
  Between 18 and 65 years | 111 | 103 | 22 | 0 | 236
  >=65 years | 14 | 18 | 2 | 0 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 52 | 12 | 1 | 125
  Male | 65 | 69 | 12 | 1 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 6 | 2 | 26
  Not Hispanic or Latino | 116 | 102 | 0 | 0 | 218
  Unknown or Not Reported | 4 | 6 | 18 | 0 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 72 | 57 | 1 | 0 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 0 | 0 | 6
  White | 43 | 51 | 11 | 2 | 107
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 12 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of Participants With Normalization Of Lactate Dehydrogenase (LDH) Levels
Description: LDH is an indicator of intravascular hemolysis that occurs in participants with paroxysmal nocturnal hemoglobinuria (PNH). A decrease in LDH from above the upper limit of normal (ULN) to below the ULN indicates reduction (improvement) in hemolysis. Normalization of LDH levels (LDH-N) was LDH levels less than or equal to 1 x ULN, from Day 29 through Day 183. The ULN for LDH is 246 U/L.
Time Frame: Day 29 through Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of study drug (ravulizumab or eculizumab) and had at least 1 efficacy assessment after the first infusion of study drug.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Ravulizumab: Participants received weight-based doses of ravulizumab ranging from 2400 to 3000 mg on Day 1. Thereafter, weight-based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Day 15 and every 8 weeks thereafter for 26 weeks.
- Eculizumab: Participants received 600 mg of eculizumab on Days 1, 8, 15, and 22, followed by 900 mg of eculizumab on Day 29 and every 2 weeks thereafter for 26 weeks.
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
proportion of participants | 0.536 [0.459 to 0.612] | 0.494 [0.417 to 0.570]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; A minimum of 142 participants were estimated to provide 80% power to demonstrate noninferiority of ravulizumab to eculizumab; Test type: Non-Inferiority — LDH-N was analyzed using a generalized estimating equation (GEE) approach. The model included the following terms: treatment group, history of transfusion (as a categorical variable based on the stratification factor levels), and baseline LDH level (as a continuous variable). Noninferiority margin was based on the lower bound of the 95% confidence interval (CI) for the odds ratio (OR) of ravulizumab versus eculizumab for LDH normalization being greater than an OR of 0.39; Odds Ratio (OR) = 1.187, 95% CI 2-sided [0.796 to 1.769]

2. Primary Outcome: Percentage Of Participants Who Achieved Transfusion Avoidance (TA)
Description: Transfusion avoidance was defined as the percentage of participants who remained transfusion free and did not require a transfusion per protocol-specified guidelines through Day 183.
Time Frame: Baseline through Day 183
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
percentage of participants | 73.6 [65.87 to 81.33] | 66.1 [57.68 to 74.55]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; A minimum of 193 participants were estimated to provide 80% power to demonstrate noninferiority of ravulizumab to eculizumab. The difference of percentages were calculated using stratified Newcombe CI method. Stratification factors were: observed stratification groups of packed red blood cells (pRBC)/whole blood units transfused in the 1 year prior to first dose of study drug and screening LDH levels; Test type: Non-Inferiority — Noninferiority margin was based on the lower bound of the 95% CI. Noninferiority margin was -20%; Treatment difference = 6.8, 95% CI 2-sided [-4.66 to 18.14] — Treatment difference was estimated for ravulizumab - eculizumab

3. Secondary Outcome: Percentage Of Participants With Breakthrough Hemolysis (BTH)
Description: Breakthrough hemolysis was defined as at least 1 new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 gram/deciliter (g/dL)], major adverse vascular event [MAVE, including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2 × ULN, after prior LDH reduction to <1.5 × ULN on therapy.
Time Frame: Baseline through Day 183
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
percentage of participants | 4.0 [0.56 to 7.44] | 10.7 [5.23 to 16.26]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; The difference of percentages was calculated using stratified Newcombe CI method. The stratification factors were: observed stratification groups of pRBC units transfused in the 1 year prior to first dose of study drug and screening LDH levels; Test type: Non-Inferiority — Noninferiority margin was based on the upper bound of the 95% CI. Noninferiority margin was 20%; Treatment difference = -6.7, 95% CI 2-sided [-14.21 to 0.18] — Treatment difference was estimated for ravulizumab - eculizumab

4. Secondary Outcome: Percent Change From Baseline In LDH Levels
Description: Baseline is defined as the average of all available assessments of LDH levels prior to first study drug dose. Estimates are based on Mixed Model for Repeated Measures (MMRM) that includes treatment group, history of transfusion (as a categorical variable based on the stratification factor levels) and baseline LDH level (as a continuous variable), study visit and study visit by treatment group interaction. An unstructured covariance structure was used.
Time Frame: Baseline, Day 183
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
percent change | -76.84 [-79.96 to -73.73] | -76.02 [-79.20 to -72.83]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; Test type: Non-Inferiority — Noninferiority margin was based on the upper bound of the 95% CI. Noninferiority margin was 20%; Treatment difference = -0.83, 95% CI 2-sided [-5.21 to 3.56] — Treatment difference was estimated for ravulizumab - eculizumab

5. Secondary Outcome: Change From Baseline In Quality Of Life As Assessed By The Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue
Description: FACIT-Fatigue score ranges from 0 to 52, with a higher score indicating less fatigue. Baseline is defined as the last non-missing value prior to first dose of study drug. Estimates are based on MMRM that includes treatment group, the observed stratification randomization indicators (history of transfusion and LDH) and baseline FACIT-Fatigue level, study visit, and study visit by treatment group interaction. An unstructured covariance structure was used.
Time Frame: Baseline, Day 183
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
units on a scale | 7.07 [5.55 to 8.60] | 6.40 [4.85 to 7.96]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; Test type: Non-Inferiority — Noninferiority margin was based on the lower bound of the 95% CI. Noninferiority margin was -5%; Treatment difference = 0.67, 95% CI 2-sided [-1.21 to 2.55] — Treatment difference was estimated for ravulizumab - eculizumab

6. Secondary Outcome: Percentage Of Participants With Stabilized Hemoglobin Levels
Description: Stabilized hemoglobin was defined as avoidance of a ≥2 g/dL decrease in hemoglobin level from baseline in the absence of transfusion through Day 183.
Time Frame: Baseline through Day 183
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab | Eculizumab
Number analyzed (Participants) | 125 | 121
percentage of participants | 68.0 [59.82 to 76.18] | 64.5 [55.93 to 72.99]
Statistical Analysis 1: Comparison: Ravulizumab vs Eculizumab; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — Noninferiority margin was based on the lower bound of the 95% CI. Noninferiority margin was -20%; Treatment difference = 2.9, 95% CI 2-sided [-8.80 to 14.64] — Treatment difference was estimated for ravulizumab - eculizumab

ADVERSE EVENTS:
Time Frame: Baseline up to Day 2045
Description: Treatment-emergent adverse events (TEAEs) reported below include TEAEs that occurred during or after first infusion of study treatment up to Day 2045 (end of study).
Groups:
- Ravulizumab: Primary Evaluation: Participants received weight-based doses of ravulizumab ranging from 2400 to 3000 mg on Day 1. Thereafter, weight-based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Day 15 and every 8 weeks thereafter for 26 weeks.
- Eculizumab: Primary Evaluation: Participants received 600 mg of eculizumab on Days 1, 8, 15, and 22, followed by 900 mg of eculizumab on Day 29 and every 2 weeks thereafter for 26 weeks.
- Ravulizumab/Ravulizumab: Extension Period; Eculizumab/Ravulizumab: Extension Period: After completion of the Primary Evaluation Period, all participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 5 years.
- Ravulizumab-Adults; Ravulizumab-Pediatrics: Participants in this group rolled over from other ongoing studies of ravulizumab intravenous in participants with PNH into the extension period of this study and received weight-based doses of ravulizumab for up to 5 years.
Arm/Group | Ravulizumab: Primary Evaluation | Eculizumab: Primary Evaluation | Ravulizumab/Ravulizumab: Extension Period | Eculizumab/Ravulizumab: Extension Period | Ravulizumab-Adults | Ravulizumab-Pediatrics
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/121 | 4/124 | 4/119 | 0/24 | 0/2
Serious Adverse Events (participants affected / at risk) | 11/125 | 9/121 | 52/124 | 43/119 | 2/24 | 0/2
Other Adverse Events (participants affected / at risk) | 87/125 | 86/121 | 102/124 | 100/119 | 13/24 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ravulizumab: Primary Evaluation (N=125) | Eculizumab: Primary Evaluation (N=121) | Ravulizumab/Ravulizumab: Extension Period (N=124) | Eculizumab/Ravulizumab: Extension Period (N=119) | Ravulizumab-Adults (N=24) | Ravulizumab-Pediatrics (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 7 | 2 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 4 | 3 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 5 | 6 | 0 | 0
Systemic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/60 | 0/52 | 1 | 1 | 0 | 0 — This is a sex-specific adverse event that only affects female participants.
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 4 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Chikungunya virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 6 | 3 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 3 | 2 | 0 | 0
Cystitis escherichia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Fungal endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Intracranial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ravulizumab: Primary Evaluation (N=125) | Eculizumab: Primary Evaluation (N=121) | Ravulizumab/Ravulizumab: Extension Period (N=124) | Eculizumab/Ravulizumab: Extension Period (N=119) | Ravulizumab-Adults (N=24) | Ravulizumab-Pediatrics (N=2)
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 10 | 12 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 14 | 13 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 10 | 8 | 11 | 0 | 0
Pyrexia (General disorders) | 6 | 11 | 22 | 18 | 2 | 0
Nasopharyngitis (Infections and infestations) | 11 | 20 | 14 | 26 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 7 | 30 | 25 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 9 | 8 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11 | 17 | 12 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 12 | 11 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 9 | 4 | 7 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 7 | 4 | 9 | 0 | 0
Headache (Nervous system disorders) | 45 | 40 | 16 | 20 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 14 | 18 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 6 | 4 | 10 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 7 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 4 | 0 | 0
Palpitations (Cardiac disorders) | 7 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 10 | 5 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 10 | 5 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 8 | 10 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 7 | 4 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 4 | 0
Chest pain (General disorders) | 0 | 0 | 8 | 3 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 5 | 10 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 7 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 19 | 16 | 9 | 0
Cystitis (Infections and infestations) | 0 | 0 | 8 | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 9 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 9 | 11 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 5 | 6 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 8 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 9 | 8 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 6 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 12 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 6 | 11 | 6 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 7 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 7 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 7 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT02946463/Prot_003.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT02946463/SAP_004.pdf